CLINICAL TRIAL: NCT03398018
Title: Efficacy of Repository Corticotropin Injection in Patients With Severe and Recalcitrant Keratoconjunctivitis Sicca
Brief Title: Repository Corticotropin Injection in Keratoconjunctivitis Sicca
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change of direction
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jason Nichols, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F00000001
Record Dates: First submitted 2018-01-02; First posted 2018-01-12 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: dry eye; corticotropin
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Treated with repository corticotropin injection
  Interventions: Drug: repository corticotropin injection

INTERVENTIONS:
Drug: repository corticotropin injection — 80 units twice per week as a subcutaneous injection
  Other Names: HP Acthar Gel

SUMMARY:
The purpose of this pilot study is to assess repository corticotropin injection (RCI) in the form of H.P. Acthar Gel in patients with severe keratoconjunctivitis sicca (KCS, or dry eye disease). This pilot study is a non-randomized, open-label, interventional study to assess the efficacy and timeline of RCI for the treatment of severe KCS recalcitrant to conventional therapy. The purpose is to acquire preliminary data to support and guide the design of a future, double-masked, randomized, controlled clinical trial.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, interventional pilot study with sixteen weeks (112 days) of active treatment, a possible twelve-week treatment extension, and twenty-four weeks of washout follow-up. Intervention is with HP Acthar Gel dosed at 80 U BIW SC indicated for use in anterior segment disease and keratitis. Data will be collected from five subjects. All subjects will be treated with 80 U BIW SC and clinically examined at two, four, six, nine, twelve, and sixteen weeks with a potential extension of up to twenty-eight weeks. Extension will be contingent upon specific outcome criteria defined in this protocol. Four clinical visits will occur at two, four, eight, and twelve weeks after initiating the drug taper to assess for regression of the signs and symptoms of KCS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe keratoconjunctivitis sicca (KCS) as defined by meeting at least three of the following in the same or both eye(s): (1) OSDI ≥ 33, (2) sum corneal staining with fluorescein of ≥ 5 in at least one eye, (3) MMP-9 concentration ≥ 40 ng/ml in at least one eye as measured by InflammaDry®, and (4) bulbar hyperemia of ≥ 2.0 in at least one eye as measured by the Oculus Keratograph® 5M
* Recalcitrant or intolerant to treatment with cyclosporine 0.05% ophthalmic emulsion (Restasis®) or lifitegrast 5% ophthalmic solution (Xiidra®)

Exclusion Criteria:

* Past or present history of: scleroderma, osteoporosis, systemic bacterial or fungal infection (including but not limited to tuberculosis), psychosis, ocular herpes simplex, peptic ulcer, congestive heart failure, diabetes mellitus, myasthenia gravis, hypothyroidism, liver cirrhosis, primary adrenocortical insufficiency or adrenocortical hyperfunction, central serous chorioretinopathy.
* Any corticosteroid use within 60 days of study enrollment
* Topical cyclosporine 0.05% ophthalmic emulsion (Restasis) or lifitegrast 5% ophthalmic solution (Xiidra) use within 60 days of study enrollment
* Recent surgery within 90 days
* Current uncontrolled, sustained hypertension
* Post-prandial blood glucose value of ≥ 140 mg/dl as measured at the baseline visit
* Sensitivity to proteins of porcine origin
* Anticipated administration of live or live attenuated vaccines during the course of the study
* Known sensitivity to steroid or complications from prior steroid use that subject is unwilling to tolerate
* Pregnancy (as assessed by urine hCG) or nursing
* Participation in a clinical trial involving a drug or device within the past 30 days
* Investigator discretion based upon medical history and/or opinion of ability to maintain protocol compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Conjunctival hyperemia | 16 weeks
  Change from baseline in bulbar conjunctival hyperemia as measured by the Oculus Keratograph 5M
Corneal staining | 16 weeks
  Change from baseline in corneal staining with fluorescein

SECONDARY OUTCOMES:
Patient symptoms | 16 weeks
  Change from baseline in patient symptoms as measured by Ocular Surface Disease Index (OSDI)
Tear cytokine concentration | 16 weeks
  Change from baseline in tear cytokine concentration as measured by Raybiotech Human Dry Eye Disease Array Q1

OTHER OUTCOMES:
Needle Fear | 16 weeks
  Change from baseline in Needle Fear Survey

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Nichols, OD, MPH, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No